CLINICAL TRIAL: NCT01576692
Title: A Safety/Feasibility Trial of the Addition of the Humanized Anti-GD2 Antibody (hu14.18K322A) With and Without Natural Killer Cells to Chemotherapy in Children and Adolescents With Recurrent/Refractory Neuroblastoma
Brief Title: Combination Chemotherapy, Monoclonal Antibody, and Natural Killer Cells in Treating Young Patients With Recurrent or Refractory Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: CURE Childhood Cancer, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GD2NK; NCI-2012-00495 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma; refractory neuroblastoma; natural killer cells
MeSH Terms: conditions — Neuroblastoma | interventions — humanized 3F8 anti-GD2 monoclonal antibody; Hu14.18K322A monoclonal antibody; Drug Therapy; Cyclophosphamide; Topotecan; Temozolomide; Irinotecan; Carboplatin; Ifosfamide; Etoposide; Cytokines; Interleukin-2; aldesleukin; sargramostim; IL32 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Participants receive humanized anti-GD2 antibody, chemotherapy, cytokines, and natural killer cells.
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Biological: Humanized anti-GD2 antibody; Drug: Chemotherapy; Other: Cytokines; Biological: Natural killer cells; Device: CliniMACS

INTERVENTIONS:
Biological: Humanized anti-GD2 antibody — A maximum of 6 courses of therapy may be given on the following schedule:
  * Courses 1, 3, and 5: Humanized anti-GD2 antibody + chemotherapy
  * Courses 2, 4, and 6: Humanized anti-GD2 antibody + chemotherapy, with or without natural killer (NK) cells (depending on availability of appropriate NK donor)
  * Humanized anti-GD2 antibody (hu14.18 K322A) dosage: 40 mg/m^2)/dose, over 4 hours daily
  * NK Cell dosage: minimum of 0.1 * 10^6 cells/kg; maximum of 400 * 10^6 CD45+ cells/kg, given once
  Other Names: Hu14.18K322A monoclonal antibody
Drug: Chemotherapy — Chemotherapy may include the following at the dosages shown below:
  * cyclophosphamide: 400 mg/m^2 IV days 1-5
  * topotecan: 1.2 mg/m^2 IV days 1-5
  * temozolomide: 150 mg/m^2 PO at least 1 hour before irinotecan
  * irinotecan: 50 mg/m^2 IV over 1 hour daily for 5 days
  * carboplatin (AUC 8-dosing based on GFR), IV day 1 only
  * ifosfamide: 2 g/m2 IV days 1-3
  * etoposide: 100 mg/m2 days 1-3
  Other Names: Cytoxan; Hycamtin; Temodar; Camptosar; Paraplatin; Ifex; VP-16; Vepesid
Other: Cytokines — Cytokines may be given at the following dosages:
  * interleukin-2: 1 million units/m^2 SQ beginning day 6 of each chemotherapy course and continued every other day for 6 doses
  * GM-CSF: 250 mcg/m^2/day beginning on day 7 or day 8 of chemotherapy course and continued daily through the nadir until ANC >2,000/mm^3
  Other Names: IL-2; Aldesleukin; Proleukin; Sargramostim; Leukine
Biological: Natural killer cells — NK cells from haploidentical family donor will be infused on day 7 or 8, depending on course. NK cells may be infused in either the inpatient or outpatient setting by a physician, Physician Assistant, Nurse Practitioner, or qualified RN. Careful monitoring and supportive care during NK cell infusion will be guided in part by the Standard Operating Procedures for Lymphocytes Infusions in the St. Jude Nursing Policy & Procedure Manual.
  Other Names: NK cells
Device: CliniMACS — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest, such as CD3+ human T cells.
  Other Names: Cell Selection System

SUMMARY:
This is a safety / feasibility trial evaluating the combination of a humanized anti-GD2 antibody (HU14.18K322A) manufactured at the Children's GMP, LLC at St. Jude with allogeneic natural killer (NK) cells and standard chemotherapy in children with relapsed or refractory neuroblastoma.

DETAILED DESCRIPTION:
Eligible participants will receive chemotherapy combined with Hu14.18K322A antibody daily for four consecutive days. Those participants who go on to receive the second course of chemotherapy with Hu14.18K322A will receive an infusion of allogeneic NK cells after the 4th dose of Hu14.18K322A antibody. A maximum of six courses will be given.

Primary Objective:

* To observe and describe the toxicities associated with humanized anti-GD2 antibody (hu14.18K322A) with and without allogeneic NK cells when given with repeated cycles of chemotherapy to children with refractory/relapsed neuroblastoma.

Secondary Objective:

* To describe response, time to progression, event-free and overall survival.
* To evaluate the feasibility of administering NK cells from a suitable donor after completion of the last dose of hu14.18K322A in three repeated cycles of chemotherapy

ELIGIBILITY:
INCLUSION CRITERIA (Participant):

* Diagnosis of recurrent or refractory neuroblastoma.
* Age < 22 years at the time of enrollment.
* Measurable or evaluable (detectable by bone scan or MIBG, but not measurable) disease.
* Organ function: Must have adequate organ and marrow function as defined by the following parameters:

  * Bone marrow: Absolute neutrophil count (ANC) > 750/mm3; Platelets > 75,000/mm3 (no platelet transfusions for at least 1 week)
  * Hepatic: Total bilirubin ≤ 2 x upper limit of normal (ULN) for age; SGPT (ALT) ≤ 2.5 x ULN for age.
  * Renal: Creatinine clearance or radioisotope GFR equal to or >70 ml/min/1.73m2 OR serum creatinine based on age as follows:

    * Age 5 years of age and under, then maximum serum creatinine 0.8 mg/dL
    * Age >5 and equal to or <10 years, then maximum serum creatinine 1.0 mg/dL
    * Age >10 and equal to or <15 years, then maximum serum creatinine 1.2 mg/dL
    * Age >15 years, then maximum serum creatinine 1.5 mg/dL
  * Cardiovascular: Shortening fraction > or equal to 27% by echocardiogram; Corrected QT interval < or equal to 450 milliseconds
* Performance status: Karnofsky > or equal to 50 for > 10 years of age; Lansky > or equal to 50 for children equal to or < 10 years of age.
* Prior therapy: Participant must have fully recovered from the acute toxic effects of all prior therapy prior to enrolling on study.

  * Myelosuppressive chemotherapy: Must not have received myelosuppressive therapy within 2 weeks prior to study entry (4 weeks if nitrosurea).
  * Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with biologic agent, including retinoic acid. At least 6 weeks must have elapsed since prior therapy that includes a monoclonal antibody. Participants receiving IVIG are eligible; however, participant must not receive IVIG during the 4 days of antibody infusion.
  * Radiation therapy: At least 2 weeks since prior local radiation therapy at the time of study entry.
  * Growth factors: Must not have received hematopoietic growth factors (G-CSF, GM-CSF) for at least 1 week prior to study entry.
  * Investigational agent: Must not have received investigational agent within 7 days of study entry.
  * Immune therapy: Must not have received immunosuppressive (including glucocorticoids), immunostimulatory or any immunomodulatory treatment within 2 weeks of study entry. Steroid containing inhalers, steroid replacement for adrenal insufficiency and steroid premedication for prevention of transfusion or imaging contrast-agent related allergic reaction will be permitted.
* Participants may have had prior CNS metastasis providing: CNS disease has been previously treated and CNS disease has been clinically stable for 4 weeks prior to study entry (assessment must be made by CT or MRI).
* Written informed consent following institutional and federal guidelines.

EXCLUSION CRITERIA (Participant):

* Prior monoclonal antibody: Participants having received in vivo monoclonal anti-GD2 antibodies for biologic therapy or for tumor imaging are ineligible if they have experienced a severe allergic reaction while receiving prior anti-GD2 therapy.
* Pregnancy or breast feeding: Study participants who are pregnant are not eligible for this study. Pregnancy tests must be obtained in girls who are > 10 years of age or post-menarchal within 7 days prior to study enrollment. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during participation in the trial. Breast feeding should be discontinued if a mother wishes to participate in this study.
* Allergy: Known hypersensitivity to other recombinant human antibodies.
* An uncontrolled infection.
* Participants who have not started protocol therapy within 7 days of study enrollment.

INCLUSION CRITERIA (Donor):

* Donor is a partially matched family member.
* Donor is HIV negative.
* Donor is at least 18 years of age.
* Donor is not pregnant.
* Donor does not have any other medical condition that, in the opinion of an independent physician, precludes performance of an apheresis procedure.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing unacceptable toxicity associated with humanized anti-GD2 antibody/chemotherapy (course 1) and anti-GD2 antibody/chemotherapy/NK cells (course 2). | First two courses of treatment (42 days)
  Unacceptable toxicities are defined as: 1) any grade 4 toxicity that does not return to baseline by day 35, 2) any toxicity requiring the use of pressors, including grade 4 acute capillary leak syndrome or grade 3 or 4 hypotension, 3) any toxicity requiring ventilation support, including grade 4 respiratory toxicity, 4) grade 4 neutropenia or thrombocytopenia lasting > 35 days (only during course 2), and 5) death from toxicity.

SECONDARY OUTCOMES:
Response to treatment | Baseline and three (3) weeks following courses 2, 4, and 6
  Clinical outcome measured as response to therapy using the RECIST response evaluation criteria in solid tumors and/or clearing of bone marrow and/or improvement in MIBG scans.
Time to progression. | Time from date of study enrollment to date of disease progression or recurrence, assessed up to 4.5 years.
Event free survival. | Time from date of study enrollment to date of first event (relapsed or progressive disease, second malignancy or death from any cause) or to the date of last contact for patients without events, assessed up to 4.5 years.
  Event-free survival will be estimated using the method of Kaplan and Meier.
Overall survival | Time from date of study enrollment to date of death from any cause or to the date of last contact for survivors, assessed up to 4.5 years.
  Survival will be estimated using the method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne L. Furman, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols